CLINICAL TRIAL: NCT03279328
Title: Evaluating Skin Appearance Following 5-Flourouracil Cream for Treatment of Actinic Keratosis and the Effects of Topical Agents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1708724736
Record Dates: First submitted 2017-09-07; First posted 2017-09-12 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Topical Steroid Ointment (Active Comparator): One side of the face will receive a Topical Steroid ointment twice daily for seven days.
  Interventions: Drug: Topical Steroid Ointment
- Vaseline (Active Comparator): One side of the face will receive Vaseline twice daily for seven days.
  Interventions: Other: Vaseline
- Skin Barrier Moisturizer (Active Comparator): One side of the face will receive Skin Barrier Moisturizer twice daily for seven days.
  Interventions: Drug: Skin Barrier Moisturier

INTERVENTIONS:
Drug: Topical Steroid Ointment — Based on randomization, the subject will either apply Topical Steroid Ointment, Vaseline or skin barrier repair moisturizer to one side of the face for seven days.
  Arms: Topical Steroid Ointment
Other: Vaseline — Based on randomization, the subject will either apply Topical Steroid Ointment, Vaseline or skin barrier repair moisturizer to one side of the face for seven days.
  Arms: Vaseline
Drug: Skin Barrier Moisturier — Based on randomization, the subject will either apply Topical Steroid Ointment, Vaseline or skin barrier repair moisturizer to one side of the face for seven days.
  Arms: Skin Barrier Moisturizer

SUMMARY:
This proposed project will be an open-label, split face, randomized controlled pilot study. Up to 60 patients with diffuse facial actinic keratosis will be enrolled in the study. The purpose of this study is to understand the change in skin appearance throughout 5-FU treatment course and to examine whether a topical corticosteroid and moisturizer can decrease severity and duration of skin inflammation after 5-FU treatment course.

DETAILED DESCRIPTION:
The purpose of this study to understand the change in skin appearance during and after the course of 5-FU cream in patients with AK, and compare how the appearance of skin inflammation changes with the use of topical corticosteroids and moisturizers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, at least 18 years of age
* Subject must have a diagnosis of actinic keratosis (at least 5 lesions on each side of the face)
* Able to comprehend and read the English language

Exclusion Criteria:

* Subjects who do not fit the inclusion criteria
* Concurrently have other inflammatory skin conditions.
* Prior known allergy to any components to of 5FU cream, topical steroid ointment or vaseline.

  • Subject who, in the opinion of the investigator, will be uncooperative or unable to comply with study procedures (i.e.: compliant with using 5-FU cream, topical corticosteroid or moisturizers
* Those that are prisoners or cognitively impaired.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Skin barrier biophysical properties | 2 hours
  Transepidermal water loss (TEWL) will be measured using hand-held, noninvasive skin barrier measuring devices (Tewameter)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona - Banner University Medicine Dermatology, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No